CLINICAL TRIAL: NCT04245774
Title: Comparing the Effects of Levobupivacaine and Bupivacaine in Anorectal Surgery Under Saddle Spinal Anesthesia
Brief Title: Comparing the Effects of Levobupivacaine and Bupivacaine in Saddle Spinal Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Asst. Prof. Hasan Ali KİRAZ, MD, Assistant professor, MD, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Thesis No: 224639
Record Dates: First submitted 2020-01-20; First posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Outpatients; General Surgery; Anorectal Disorder; Anesthesia; Drug Effect
Keywords: Saddle block; Hyperbaric levobupivacaine and bupivacaine; Outpatient anorectal surgery
MeSH Terms: conditions — Rectal Diseases | interventions — Levobupivacaine; Solutions; Glucose; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Participants were divided into two groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study was a double blind research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group L (Hyperbaric Levobupivacaine) (Experimental): 7,5 mg (1.5 mL) of 0,5% hyperbaric levobupivacaine injected into the intrathecal space in sitting position through L4-L5 or L5-S1 intervertebral space in 30 seconds.
  In order to obtain hyperbaric levobupivacaine, 1 mL 0.75% isobaric levobupivacaine (Chirocaine® 75 mg/10mL ampoule Abbott/Turkey, Nycomed Pharma/Norway) was added to 0.24 mL 50% Dextrose (dextrose 120 mg) (Eczacıbaşı/Turkey) and 0.26 mL distilled water.
  Interventions: Drug: Levobupivacaine (as Levobupivacaine Hydrochloride) 75 Mg/10 mL Solution for Injection Ampoule
- Group B (Hyperbaric Bupivacaine) (Active Comparator): 7,5 mg (1.5 mL) of 0,5% hyperbaric bupivacaine (Marcaine® Spinal Heavy, 0.5%, 4 mL ampoule, AstraZeneca/England, Eczacıbaşı/Turkey, dextrose content 80 mg/mL) injected into the intrathecal space in sitting position through L4-L5 or L5-S1 intervertebral space in 30 seconds.
  Interventions: Drug: Bupivacaine/Dextrose

INTERVENTIONS:
Drug: Levobupivacaine (as Levobupivacaine Hydrochloride) 75 Mg/10 mL Solution for Injection Ampoule — 7,5 mg (1.5 mL) of 0,5% hyperbaric levobupivacaine (1 mL 0.75% isobaric levobupivacaine (Chirocaine® 75 mg/10mL ampoule Abbott/Turkey, Nycomed Pharma/Norway) plus 0.24 mL 50% Dextrose (dextrose 120 mg) (Eczacıbaşı/Turkey) and 0.26 mL distilled water) injected into the intrathecal space in sitting position through L4-L5 or L5-S1 intervertebral space in 30 seconds. All patients kept in sitting position for 5 minutes with aid after intrathecal injection and than layed in supine position, finally they positioned in prone jack-knife.
  Other Names: 1 mL 0.75% isobaric levobupivacaine (Chirocaine® 75 mg/10mL ampoule Abbott/Turkey, Nycomed Pharma/Norway) plus 0.24 mL 50% Dextrose (dextrose 120 mg) (Eczacıbaşı/Turkey) and 0.26 mL distilled water.
  Arms: Group L (Hyperbaric Levobupivacaine)
Drug: Bupivacaine/Dextrose — 7,5 mg (1.5 mL) of 0,5% hyperbaric bupivacaine (dextrose content 80 mg/mL) injected into the intrathecal space in sitting position through L4-L5 or L5-S1 intervertebral space in 30 seconds. All patients kept in sitting position for 5 minutes with aid after intrathecal injection and than layed in supine position, finally they positioned in prone jack-knife.
  Other Names: Marcaine® Spinal Heavy, 0.5%, 4 mL ampoule, AstraZeneca/England, Eczacıbaşı/Turkey, dextrose content 80 mg/mL.
  Arms: Group B (Hyperbaric Bupivacaine)

SUMMARY:
İn this study; it was aimed to investigate the effects of equipotent doses of hyperbaric bupivacaine and hyperbaric levobupivacaine in outpatient anorectal surgery under saddle block. Sixty patients between the age of 18- 50 and in the risk group of ASA I-II included in the study. 7,5 mg of 0,5% hyperbaric bupivacaine or 7,5 mg of 0,5% hyperbaric levobupivacaine injected into the intrathecal space in sitting position through L4-L5 or L5-S1 intervertebral space in 30 seconds. All patients kept in sitting position for 5 minutes with aid after intrathecal injection and than layed in supine position, finally they positioned in prone jack-knife. Hemodynamic parameters like NIBP, HR, SpO2, sensory and motor block characteristics, duration of analgesia, time of first voiding, mobilization time, patient and surgeon satisfaction, adverse effects and discharge time were recorded during and after surgery.

DETAILED DESCRIPTION:
This study was completed in the General Surgery operating room within the Department of Anesthesiology and Reanimation in Gazi University Faculty of Medicine after receiving permission from Gazi University, Faculty of Medicine Local Ethics Committee (dated 28.05.2007, numbered 172). After receiving informed consent forms, the study included 60 patients aged 18-50 years in ASA I-II risk group with planned elective anorectal surgery. Those with known hypersensitivity to amid-type local anesthetics, who did not accept regional anesthesia administration, with preoperative motor and sensory loss, who did not accept participation in the study and with contraindications for spinal anesthesia method were not included in the study.

Patients did not have premedication before the operation. Patients were divided into two groups with Group B given 7.5 mg (1.5 mL) hyperbaric bupivacaine (Marcaine® Spinal Heavy, 0.5%, 4 mL ampoule, AstraZeneca/England, Eczacıbaşı/Turkey, dextrose content 80 mg/mL), while Group L were administered 7.5 mg (1.5 mL) hyperbaric levobupivacaine. In order to obtain hyperbaric levobupivacaine, 1 mL 0.75% isobaric levobupivacaine (Chirocaine® 75 mg/10mL ampoule Abbott/Turkey, Nycomed Pharma/Norway) was added to 0.24 mL 50% Dextrose (dextrose 120 mg) (Eczacıbaşı/Turkey) and 0.26 mL distilled water. While mixing hyperbaric levobupivacaine, in order to obtain accurate doses of levobupivacaine, it was measured with 50% dextrose and 1 mL distilled water in an insulin injector. The hyperbaric bupivacaine and hyperbaric levobupivacaine had specific gravity values measured in Gazi University, Central Biochemistry Laboratory (solutions were heated before measurements and set with an electronic thermometer - Microlife gold-tipped thermometer MT 3001, importer Trimpeks - İstanbul, Made in P.R.C.) at 37 ºC as 1.026 (URISYS 2400, Serial No:1744-017 part No:614-0010, Roche Diagnostics Germany, Made in Japan Production year 2005). Based on specific gravity, mean density in water at 37 ºC was accepted as 0.993 g/mL (51,72) and we calculated the solution density used in our study as 1.0188 g/mL (1.026 x 0.993 g/mL = 1.0188 g/mL).

Local anesthetics to be used for spinal anesthesia were prepared by another anesthesiologist so the researcher who would administer and monitor the patient, and the patient, did not know which was used. Sixty patients had the random double-blind study method applied according to order until each group contained 30 patients. Before administering spinal anesthesia, IV cannulation was performed on the nondominant hand with an 18-gauge (G) branule and patients were administered 8-10 mL/kg Ringer lactate solution over 10-15 minutes. The fluid amounts before anesthesia and in total were recorded. Patients taken to the operating room had ECG (II derivation), SpO2, and noninvasive blood pressure (NIBP) monitoring performed (NIHON KOHDEN, Model: BSM4113K, SN:01236, 2004 - Japan). The 4 L/min O2began to be administered through a mask and basal hemodynamic parameters for patients with preoperative motor and sensory examination were recorded as control values on the monitoring form prepared for the study.

All patients had spinal anesthesia performed in the sitting position in the L4-5 or L5-S1 interspinous space. The number of spinal puncture attempts and the successful interval were recorded. If puncture was unsuccessful on the third attempt, the case was excluded from the study. All drugs were prepared for single use under sterile conditions.

After necessary skin disinfection, the interval for the intervention had local anesthesia provided by 2 mL 2% lidocaine administered with a 22 G fine needle to infiltrate the ligamentum flavum from the skin. The appropriate interval first had a 20 G 35 mm needle introducer (guide needle) inserted from the spinal needle set. Within the introducer, a 26 G atraumatic spinal needle (Atraucan®, B.Braun, Melsungen AG) was inserted parallel to the dura fibers on the midline until the dura was passed and then the chuck of the spinal needle was removed and after clear cerebrospinal fluid (CSF) was observed the needle opening was turned toward sacral. For Group B 7.5 mg hyperbaric bupivacaine (1.5 mL) and for Group L 7.5 mg (1.5 mL) hyperbaric levobupivacaine was administered into the intrathecal space over 30 seconds and the end of drug administration was accepted as 0 minutes. Supported by an assistant, the patients were left in sitting position for 5 min and then laid supine. The break region of the operating table was placed equivalent to the iliac crista of the patient and they were given the prone jack-knife position.

Spinal anesthesia sensory block level, motor block degree and hemodynamic markers of heart rate (HR), systolic arterial pressure (SAP), diastolic arterial pressure (DAP), mean arterial pressure (MAP) and SpO2values were recorded every 2.5 min until 15 min after spinal anesthesia and later every 5 min until the end of surgery. Sensory block level was assessed using a blunt-tipped needle with the 'pin prick' test by touching appropriate dermatome on the standard dermatome map; sympathetic block degree was measured with the feeling of temperature on the skin by touching with cold alcohol sponge; and motor block level was assessed with the modified Bromage scale (0= no paralysis, thighs, legs and feet can be raised, 1= thighs cannot be moved, knees moved, 2= knees cannot be moved, ankles can be moved, 3= lower extremities cannot be moved). After identifying that all sacral dermatome could not feel the tip of the needle, the operation was allowed to begin. The duration from puncture to beginning of operation was recorded. With the 'pin prick' test, the region of surgery was checked for sufficient sensory block for analgesia. Sensory block was recorded and evaluated as the duration sensory block continued before regression to two dermatome. Sensory and motor block assessments were performed during the operation. The duration to form sufficient anesthesia for the relevant surgery, time when maximum levels were reached, maximum level, time for sensory block to regress two segments and end time for sensory block were recorded. For motor block, maximum motor block degree and formation duration, and end time for motor block were assessed and recorded. If sufficient anesthesia was not provided 20 min after administration of spinal anesthesia, the case was excluded from the study and general anesthesia was planned. MAP falling more than 20% according to control values or below 60 mmHg was accepted as hypotension, and rapid fluid replacement began (50 mL/min). If there was no response within three minutes, IV bolus 5 mg ephedrine (Ephedrine HCl ampoule, 0.05 g, 1 mL OSEL/İstanbul) was administered and total ephedrine amounts before being sent to the ward were recorded. If HR fell below 50 beats/min, it was evaluated as bradycardia and IV bolus 0.5 mg atropine (atropine sulfate, ½ mg, 1 mL ampoule, OSEL/İstanbul) was administered and it was recorded on the monitoring form.

Patients were monitored for side effects like hypotension, bradycardia, nausea, vomiting, pain, shivering, discomfort and respiratory depression during the operation and complications were recorded. At the end of surgery, total surgical duration was recorded and patient and surgical team were asked whether they were satisfied with the anesthesia method. Degree of satisfaction was recorded on a 5-point scale as 0 poor, 1 mediocre, 2 good, 3 very good and 4 perfect.

At the end of the surgical intervention, cases were placed in supine horizontal position and taken to the recovery room. In the recovery room, patients had the verbal numerical scale (VNS) explained (0= no pain, 10= most severe pain possible) and severity of pain was recorded. Patients with VNS scores above 4 were administered pethidine (Aldolan® ampoule, Pethidine HCl 100 mg/2mL Liba/İstanbul, Gerot Pharmazeutika/Austria) IM 1 mg/kg. The time for first analgesic requirements was recorded (total analgesia duration). In the first hour in the recovery room, HR, SAP, DAP, MAP, SPO2, sensory block and motor block levels were recorded every 10 minutes. Patients with normal parameters in the recovery room were sent to the general surgery ward. SAP, DAP, MAP, sensory block levels, motor block degree and side effects were recorded on the patient monitoring form prepared for the study in the ward every 30 min from the 90th minute to 3 hours and every hour from 3rd to 6th hours and at the 8th, 10th, 16th and 24th hours. Patients were requested to report their time of first urination and time of first walking on the ward. Patients without pain during postoperative monitoring in the recovery room were requested to note the time for first analgesic requirements (total analgesia duration) and wards were visited to record this information. Patients were monitored in terms of complications like headache, back ache, urinary retention, pain in legs, weakness, urinary or anal incontinence, nausea, vomiting, hypotension, and bradycardia from after the operation until discharge. Discharge day was recorded. After discharge, they were told to inform the researchers of any problems and were telephoned and monitored for headache and temporary neurologic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II risk group with planned elective anorectal surgery
* Approved to participate in the study and spinal anesthesia

Exclusion Criteria:

* Known hypersensitivity to amid-type local anesthetics
* Not to accept regional anesthesia administration
* With preoperative motor and sensory loss
* Not to accept participation in the study
* Contraindications for spinal anesthesia method

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-11-21 (Actual); Primary Completion 2008-08-13 (Actual); Study Completion 2008-12-17 (Actual)

PRIMARY OUTCOMES:
Adequate level of anesthesia for surgery | The first 20 minutes after administering spinal anesthesia.
  The time until the needle tip is not felt in all sacral dermatomes with "pin prick" test at determined time intervals after spinal anesthesia.
Time to obtain maximum sensory block | Time from administering spinal anesthesia to the end of the surgery (minutes).
  The time which the highest level of dermatome is formed when the needle tip is not felt with the "pin prick" test at the specified time intervals.
The highest level of sensory block | The maximum sensory block level reached until the end of the surgery.
  The highest dermatome level where the needle tip is not felt pointed with the "pin prick" test at the specified time intervals.
Two segment regression time of sensory block | Up to 1 hour.
  The time from the maximum sensory block level obtained to two segment regression
The end time of sensory block | First 24 hours in postoperative period.
  The time from sensory block start time until sensory block is removed in all dermatomes assessed by pin prick test.
The degree of maximum motor block | Up to 1 hour.
  With 3 points in modified Bromage score (3= lower extremities cannot be moved).
The time to obtain maximum motor block degree | Up to 1 hour.
  The time until the maximum level of motor block with 3 points in modified Bromage score (3= lower extremities cannot be moved) after spinal anesthesia.
The end time of motor block | Up to 4 hours.
  Time from motor block start time until the modified Bromage score returns to 0 again.

SECONDARY OUTCOMES:
Heart rate | From entry time to operating room until postoperative first 24 hours (minutes).
  Heart rate as beats/minute
Systolic arterial pressure | From entry time to operating room until postoperative first 24 hours (minutes).
  Non-invasive measurement of systolic arterial pressure (mmHg)
Diastolic arterial pressure | From entry time to operating room until postoperative first 24 hours (minutes).
  Non-invasive measurement of diastolic arterial pressure (mmHg)
Mean arterial pressure | From entry time to operating room until postoperative first 24 hours (minutes).
  Non-invasive measurement of mean arterial pressure (mmHg). To calculate a mean arterial pressure, double the diastolic blood pressure and add the sum to the systolic blood pressure. Then divide by 3.
Peripheral oxygen saturation - SpO2 | From entry time to operating room until postoperative first 1 hour (minutes).
  Non-invasive measurement of SpO2 (%).
First analgesic requirement | Up to 12 hours.
  The time that severity of pain measured using Verbal Numerical Scale (0= no pain, 10= most severe pain possible) above 4 points.
First mobilization time | Up to 6 hours.
  The first time the patient can mobilize in postoperative period
First voiding time | Up to 12 hours.
  The first time the patient can urinate in postoperative period
Patient satisfaction | Postoperative first 24 hours.
  Degree of satisfaction was recorded on a 5-point scale as 0 poor, 1 fair, 2 good, 3 very good and 4 perfect.
Surgeon satisfaction | Postoperative first 24 hours.
  Degree of satisfaction was recorded on a 5-point scale as 0 poor, 1 fair, 2 good, 3 very good and 4 perfect.

OTHER OUTCOMES:
Perioperative hypotension, bradycardia, nausea, vomiting and respiratory depression | From entry time to operating room until postoperative first 1 hour (minutes).
  Perioperative side effects
Postoperative hypotension, bradycardia, nausea, vomiting, respiratory depression, headache, urinary retention, back pain | Postoperative first 24 hours.
  Postoperative side effects
Number of patients with perioperative ephedrine administered. | From entry time to operating room until postoperative first 1 hour (minutes).
  The mean arterial pressure falling more than 20% according to control values or below 60 mmHg was accepted as hypotension, and rapid fluid replacement began (50 mL/min). If there was no response within three minutes, IV bolus 5 mg ephedrine was administered.
Number of patients with perioperative atropine administered. | From entry time to operating room until postoperative first 1 hour (minutes).
  If heart rate fell below 50 beats/min, it was evaluated as bradycardia and intravenous bolus 0.5 mg atropine was administered.
Number of patients discharged on operation day. | The day of the surgical operation done.
  Number of patients discharged on operation day.
Number of patients discharged on the day after operation. | One day after the day of the surgical operation done.
  Number of patients discharged on the day after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Cengiz B DEMİREL, 1, Study Director — Gazi University (formerly)

IPD SHARING:
Plan to Share IPD: No